CLINICAL TRIAL: NCT05682417
Title: Impact of Body Schema Distortion on Remission and Weight Regain in Anorexia Nervosa
Acronym: SCAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_1364
Record Dates: First submitted 2023-01-04; First posted 2023-01-12 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Body image; Body distortion
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with anorexia nervosa according to DSM-5 (Experimental): Patients over 15 years old, suffering from anorexia nervosa according to DSM-V with a BMI<18.5 and without psychiatric comorbidities
  Interventions: Device: Body Map Assessment Tool: MOVE Tool; Other: PAQ questionnaire; Other: F-DFlex questionnaire; Other: BSQ questionnaire; Other: Silhouette testing; Other: Eating Disorder Inventory - 2; Other: EDEQ questionnaire; Other: STAI questionnaire; Other: BECK questionnaire

INTERVENTIONS:
Device: Body Map Assessment Tool: MOVE Tool — In VR, a spherical object approaches with linear trajectory the body of patients, it can be sent to 4 parts of the body (mid-arm/waist/hip/mid-thigh) both left and right side. Several conditions are presented, either the trajectory leads the object to touch the body, or it passes at ≠ distances from it. Patient is instructed to move only if he thinks the object will touch his body.
  Procedure begins with a measurement taken on 3 body locations via the Move tool (shoulders/hips/thighs) to create an avatar allowing the tool to determine whether or not movement was necessary. Then, the movement of the patient is recorded. For each object/body distance, the software determines if dodging was necessary. The overestimation of the body schema corresponds to the average distance from which the patient considers that the object would have touched her body and performs a dodging movement, compared to her real morphological dimensions. This generates a body limit distortion % for each body area.
Other: PAQ questionnaire — This questionnaire has been translated and validated (French version, Luminet et al., 2021). This is a self-reported measure of alexithymia in 24 items. It is designed to measure all the components of alexithymia for both negative and positive emotions. Five subscale scores and six composite scores can be obtained from the questionnaire, with high scores indicating higher levels of alexithymia.
Other: F-DFlex questionnaire — This questionnaire (Detail and Flexibility Questionnaire, French version of Maria et al, 2020) assesses cognitive rigidity. This questionnaire assesses two frequently impaired cognitive dimensions in people with anorexia nervosa, central coherence and cognitive flexibility in daily functioning using 20 self-completed items.
Other: BSQ questionnaire — The Body Shape Questionnaire (BSQ, translated and validated in French by Rousseau et al., 2005) is a one-dimensional Anglo-Saxon self-questionnaire of 34 items that assesses concerns about body shape over the past four weeks. Responses are scored on a 6-point Likert scale. A score of 1 ("never") means the problem is not present, up to a score of 6 ("always") which means the problem is always present. The higher the score, the more the concern/dissatisfaction with one's body tends to be pathological.
Other: Silhouette testing — Body overestimation is assessed by the computerized silhouette test (adapted from Gardner & Brown, 2010, Van der Linder et al., 2017). Twenty-seven Body Mass Index silhouettes ranging from 11 to 40 are presented to participants in random order. For each silhouette presented, the participant answers whether or not the silhouette presented corresponds to her current silhouette. A body underestimation index is calculated as follows: Estimated figure average BMI - actual BMI.
Other: Eating Disorder Inventory - 2 — Allows self-assessment of symptoms of eating disorders. It is composed of 91 questions grouped into 11 subscales that assess specific cognitive and behavioral dimensions: desire for thinness, bulimia, body dissatisfaction, feeling of inefficiency, perfectionism, interpersonal distrust, interoceptive sensitivity, fears relating to maturity, asceticism. , impulsiveness and social insecurity. For each item, participants can answer "always", "usually", "often", "sometimes", "rarely" or "never". The score for each item is between 0 and 3. The subscale scores are calculated by simply adding all the item scores for each specific subscale. This questionnaire has demonstrated good internal consistency, test-retest reliability, and validity (Garner, 1991)
Other: EDEQ questionnaire — Or "Eating Disorders Examination - Questionnaire" (Fairburn & Beglin, 2008). This questionnaire assesses eating behaviors and concerns about weight and body shape, using 28 items focusing on these aspects over the past 28 days.
Other: STAI questionnaire — The Spielberger Anxiety Scale (STAI) State and Trait. This questionnaire includes two distinct scales: one evaluating the current state of anxiety (STAI form Y-A: feelings of apprehension, tension, nervousness and worry that the subject feels at a precise precise moment) and the second evaluating the anxious personality trait (STAI form Y-B: feelings of apprehension, tension, nervousness, and worry that the subject usually feels). The Y version was developed in order to eliminate the items having appeal to depression compared to the initial form. Each scale has 20 items. This questionnaire has good psychometric qualities regarding validity, reproducibility and inter-individual sensitivity. It correlates well with other anxiety questionnaires in a literature review of anxiety questionnaires (Elwood, 2012).
Other: BECK questionnaire — Beck Depression Inventory (Beck, 1987). The inventory is composed of items related to depressive symptoms as well as physical symptoms. This is a questionnaire that gives a quantitative estimate of the intensity of depression. Investigators will use the abbreviated version consisting of 13 items, each item comprising 4 sentences corresponding to 4 degrees of increasing intensity of a symptom on a scale of 0 to 3. The total score corresponds to the sum of the different items and makes it possible to judge the presence of depression and its intensity.

SUMMARY:
Anorexia nervosa is a predominantly female eating disorder that most often appears in adolescence. The latter leads to strict and voluntary food deprivation for several months or even years. The lifetime prevalence of anorexia is 1.4% in women and 0.2% in men.

Ultimately, only half of people treated for anorexia nervosa in adolescence recover, 30% simply improve, 21% suffer from chronic disorders and 5 to 6% die. At the same time, between a quarter and half of patients abandon their current treatment, including during hospitalization. Relapses occur during the evolution of anorexia nervosa. Even more worrying, mortality is highest the year following the patient's discharge from hospital. This appears to be due to somatic complications in more than half of cases (most often cardiac arrest), to suicide in 27% of cases.

Researchers are still trying to clarify the mechanisms involved in the emergence and persistence of this disorder. The objective is to obtain more verified and faster cures. However, the obstacles to successful treatment are mainly due to the denial of disorders and thinness.

From a neurocognitive perspective, the representation one has of one's body is underpinned by two types of representations, i.e. body image and body schema.

It has long been shown that body image is altered in anorexia nervosa. More recently, authors have shown that the distortion of the body representation was however more extensive and also affected the body schema. Patients find themselves too fat despite obvious thinness and move through space as if this were really the case.

Worryingly, these distortions in bodyschema seem to persist after therapeutic management. Despite the potential role of body-scheme distortions in maintaining the disorder, as well as the risk of relapse, the difficulties in assessing body-scheme are significant. Indeed, recovery in these pathologies is often determined according to the Body Mass Index, self-declaration and questionnaires evaluating body image, again limiting the verification of the resorption of distortions in the body schema.

Investigators have therefore developed the systematic, ergonomic and simplified evaluation of the body schema in patients suffering from anorexia nervosa at the time of diagnosis in an expert center, but also during follow-up evaluations thanks to the use of an evaluation platform of the body schema, i.e. the body in brain platform, developed by the LIP/PC2S laboratory and the SATT Linksium which allows the evaluation of the body schema.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 15 years old
* Women
* Patient with a BMI <18.5
* Patient suffering from anorexia nervosa (DSM V, 2013)
* Patient agreeing to participate in the study with signed informed consent (Or whose parents/holder of parental authority have signed the informed consent)
* Patient affiliated to a Social Security plan or beneficiary of such a plan

Exclusion Criteria:

* Adult patients protected by a legal protection measure (guardianship, curatorship, etc.)
* Patients participating in another research that may interfere with this research
* Patients with acute and co-occurring psychiatric comorbidities (suicidal crisis, delusions)
* Patients not fluent in French
* Pregnant, parturient or breastfeeding women (on questioning of the patient)
* Persons deprived of their liberty by a judicial or administrative decision
* Persons admitted to a health or social establishment for purposes other than research
* Patients with any current pathology or history of psychotic disorders, migraine, epilepsy, balance disorders, vertigo, visual disorders, proprioceptive disorders and/or neuromuscular disorders.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Overestimation of the body schema | Baseline (T0); 6 months after baseline (T+6); 12 months after baseline (T+12)
  Overestimation of the body schema (in percentage) assessed by the body schema assessment platform (MOVE tool, motion assessment in virtual reality).
  Overestimation of the body schema (percentage of distortion) will be compared to normal values, and then compared with the percentages at T+6 and T+12.

SECONDARY OUTCOMES:
Weight/height ratio, expressed by body mass index (BMI) | Baseline T0; 6 months; 12 months
  This weight(kg)/height(m)2 ratio is measured using a mathematical formula. It will be analyzed using the DSM-V reference table to measure the severity of the disorder.
  Lightweight: BMI > or = 17 kg/m2 Moderate: BMI 16-16.99 kg/m2 Severe: BMI: 15-15.99 kg/m2 Extreme: BMI < 17 kg/m2
Body overstatement | Baseline T0; 6 months; 12 months
  Body overestimation is assessed using the computerized silhouette test. This test presents 27 figures with BMIs ranging from 11 to 40. The patient answers whether or not the figure presented corresponds to his current figure.
Alexithymia score | Baseline T0; 6 months; 12 months
  Alexithymia is assessed with the PAQ questionnaire consisting of 24 questions with 7 degrees of response. (1 strongly disagree - 2 - 3 - 4 Neither agree nor disagree -5 - 6 - 7 strongly agree)
Cognitive rigidity score | Baseline T0; 6 months; 12 months
  The cognitive rigidity score is measured with the D-Flex questionnaire comprising 20 questions. The patient must then respond to the proposed statements using a 6-point scale (Strongly disagree (1), Somewhat disagree (2), Somewhat disagree (3), Somewhat agree (4) , Somewhat agree (5, Strongly agree (6).
Body dissatisfaction score | Baseline T0; 6 months; 12 months
  Body dissatisfaction is measured with the BSQ questionnaire comprising 34 questions rated from 1 (never) to 6 (Always)
Eating behavior assessed by the EDI-2 questionnaire | Baseline T0; 6 months; 12 months
  The eating behavior will be assessed by the EDI-2 questionnaire
Eating behavior assessed by the EDE-Q questionnaire | Baseline T0; 6 months; 12 months
  The eating behavior will be assessed by the EDE-Q
Level of anxiety | Baseline T0; 6 months; 12 months
  Anxiety is measured by STAI questionnaire.
Level of Depression | Baseline T0; 6 months; 12 months
  Depression is measured by BECK questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Referral Center for Eating Disorders. Neurological Hospital-GH East / Hôpital Neurologique Pierre Wertheimer GHE HCL, Bron, France

IPD SHARING:
Plan to Share IPD: No